CLINICAL TRIAL: NCT00686205
Title: Evaluation of a Human Immunodeficiency Virus (HIV) Blood Screening Assay
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 7B5-02-05R05
Record Dates: First submitted 2008-05-21; First posted 2008-05-29 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-12

CONDITIONS: Healthy Donors; HIV Positive
Keywords: healthy donors; HIV positives
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABBOTT PRISM HIV O Plus assay for Specificity (Experimental): All subjects will have their blood tested by the investigational HIV test.
  Interventions: Device: collection of follow-up sample based on PRISM HIV O Plus result
- ABBOTT PRISM HIV O Plus Assay for Sensitivity (No Intervention): Samples collected from specimen vendors or from specimen collection studies were tested by the investigational HIV assay.

INTERVENTIONS:
Device: collection of follow-up sample based on PRISM HIV O Plus result — Test blood samples with investigational HIV assay. If results are reactive, donors may be deferred and asked to return for a follow-up blood draw.
  Arms: ABBOTT PRISM HIV O Plus assay for Specificity

SUMMARY:
To test blood samples from volunteer donors of whole blood and blood components using a new investigational test that detects human immunodeficiency virus (HIV) infection. Results will be compared to the current HIV screening assay.

ELIGIBILITY:
Inclusion Criteria:

* Healthy donors that have consented to study

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24111 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Mississippi Valley Regional Blood Center, Davenport, Iowa
  - Community Blood Center of Greater Kansas City, Kansas City, Missouri
  - Community Blood Center, Dayton, Ohio
  - American Red Cross, Philadelphia, Pennsylvania
  - Interstate Blood Bank, Inc., Memphis, Tennessee
  - South Texas Blood And Tissue Center, San Antonio, Texas
  - Puget Sound Blood Center, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21606 donors enrolled from 6 geographically distinct blood donor and 1 plasmapheresis center. All donors were eligible if they signed a study consent form.
  In addition, 1388 specimens positive for HIV antibodies and 1117 specimens from US individuals at increased risk of HIV infection or from an HIV-2 endemic area.
Pre-assignment Details: All subjects were assigned to one group. There was no pre-screening criteria specific for this study.
Groups:
- ABBOTT PRISM® HIV O Plus Assay Results for Specificity: Blood specimens collected from donors were tested by the investigational HIV test.
- ABBOTT PRISM® HIV O Plus Assay Results for Sensitivity: Samples collected from specimen vendors or from specimen collection studies were tested by the investigational HIV assay.
Period: Overall Study
Arm/Group | ABBOTT PRISM® HIV O Plus Assay Results for Specificity | ABBOTT PRISM® HIV O Plus Assay Results for Sensitivity
Started | 21606 | 2505
Completed | 15599 | 1524
Not Completed | 6007 | 981
Not completed — Protocol Violation | 127 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Specimen handling procedure altered | 5878 | 0
Not completed — Specimens not confirmed HIV positive | 0 | 981

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABBOTT PRISM® HIV O Plus Assay Results for Specificity | ABBOTT PRISM® HIV O Plus Assay Results for Sensitivity | Total
Number analyzed (Participants) | 21606 | 2505 | 24111
Age, Customized [Number; unit: Participants]
  >= 17 years | 21606 | 2454 | 24060
  not collected | 0 | 51 | 51
Sex/Gender, Customized [Number; unit: Participants]
  Male | 0 | 1683 | 1683
  Female | 0 | 441 | 441
  Not Collected | 21606 | 381 | 21987
Region of Enrollment [Number; unit: participants]
  United States | 21606 | 1614 | 23220
  Côte D'Ivoire | 0 | 840 | 840
  Cameroon | 0 | 51 | 51

OUTCOME MEASURES:

1. Primary Outcome: PRISM HIV O Plus Test Data for Specificity
Description: Negative HIV status was determined by the results of the HIV-1/HIV-2 comparator assay and HIV-1 qualitatitve RNA.
Time Frame: 12 months
Population: The analysis was per the protocol.
Measure: Number; unit: participants
Groups:
- HIV Negative Donors: Donors with HIV-1/2 negative results using reference test and negative by HIV-1 RNA test
Arm/Group | HIV Negative Donors
Number analyzed (Participants) | 15599
participants
  PRISM HIV O Plus reactive | 10
  PRISM HIV O Plus nonreactive | 15589
Statistical Analysis 1: Comparison: HIV Negative Donors; Test type: Superiority or Other; Binomial Exact; Sample size is based on power of 80%, alpha level of 0.05, using the binomial distribution when comparing to a lower bound of specificity at 99.84; Clinical Specificity = 99.94, 95% CI [99.88 to 99.97]

2. Primary Outcome: PRISM HIV O Plus Test Data for Sensitivity
Description: Final HIV status was determined according to a supplemental testing algorithm for specimens positive by the investigational assay. Supplemental testing involved HIV-1 Western blot, HIV-2 EIA, HIV-2 Western blot and HIV-1 ribonucleic acid (RNA).
Time Frame: 12 months
Population: 1,388 specimens from individuals positive for HIV antibodies and 136 specimens positive by supplemental testing from US individuals at increased risk of HIV infection or from an HIV-2 endemic area. These 1,524 specimens were used for the sensitivity calculation.
Measure: Number; unit: participants
Groups:
- HIV Positive Samples: Known HIV-1 or HIV-2 positive samples were used. Samples were determined to be positive by HIV-1 or HIV-2 western blot.
Arm/Group | HIV Positive Samples
Number analyzed (Participants) | 1524
participants
  PRISM HIV O Plus reactive | 1524
  PRISM HIV O Plus nonreactive | 0
Statistical Analysis 1: Comparison: HIV Positive Samples; Test type: Superiority or Other; Binomial Exact; Clinical Sensitivity = 100.00, 95% CI [99.76 to 100.00]

ADVERSE EVENTS:
Time Frame: Subject related adverse events related to blood collection of the 19 follow-up specimens - 8/23/07 to 8/12/08.
Description: Adverse event reporting was only applicable to the 19 donors that returned for follow-up specimen collection. Adverse event reporting does not apply to the donor specimens collected as part of the routine donation or for the specimens used for sensitivity provided by Abbott.
  There were no device adverse events associated with testing.
Arm/Group | ABBOTT PRISM® HIV O Plus Assay Results for Specificity | ABBOTT PRISM® HIV O Plus Assay Results for Sensitivity
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/0
Other Adverse Events (participants affected / at risk) | 0/19 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must provide a copy of any proposed publication or presentation at least 30 days prior to submission for sponsor's review/approval. The PI must incorporate changes as the sponsor requires in order to protect the sponsor's proprietary rights and interests. The sponsor may require the PI to include acknowledgement of the sponsor's role in the study. The PI may be requested to delay publication/presentation an extra 60 days to enable sponsor to secure patent or other proprietary protection.